CLINICAL TRIAL: NCT04748172
Title: The Effect of COVID -19 mRNA Vaccine on Ovarian Reserve
Brief Title: COVID-19 Vaccine and Ovarian Reserve
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Aya Mohr-Sasson, Principal Investigator, Sheba Medical Center
Other Study IDs: 8121-21-SMC
Record Dates: First submitted 2021-02-06; First posted 2021-02-10 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Fertility Issues; Vaccine Adverse Reaction
Keywords: Ovarian reserve; Corona-19 virus; SARS-CoV-2
MeSH Terms: conditions — Infertility | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples evaluated for Anti Mullarian Hormone (AMH)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Women who are planning to be vaccinated: Women that are planning to be vaccinated, before receiving the first shot of the vaccine
  Interventions: Biological: SARS-CoV-2 virus vaccines; Diagnostic Test: AMH sampling; Diagnostic Test: anti Covid-19 antibody levels (Serology)

INTERVENTIONS:
Biological: SARS-CoV-2 virus vaccines — mRNA SARS-CoV-2 virus vaccines ( By Pfizer or Moderna)
Diagnostic Test: AMH sampling — Blood sample for AMH on recruitment and after three months
Diagnostic Test: anti Covid-19 antibody levels (Serology) — Blood sample for IgG against S1 protein after three months

SUMMARY:
As Israel is the first country to widely vaccinate its population using the mRNA vaccine against COVID-19, evaluating its influence on ovarian reserve is essential .

DETAILED DESCRIPTION:
Introduction:

Although there is as yet no scientific evidence that a SARS-CoV-2 virus infection could have negative effects on fertility, currently the possibility that the virus could affect sperm function and egg performance cannot be excluded. Previous studies have already shown an association between influenza and infertility. SARS-CoV-2 seems to be far more aggressive in terms of severe illness, morbidity and mortality in comparison to common influenzas, thus it is reasonable to hypothesize a possible substantial effect of Covid-19 on fertility.

At the cellular level, common influenza viruses promote oxidant-sensitive pathways, leading to increased oxidative stress. This mechanism has been blamed to cause male infertility through a reduction of progressive motility in spermatozoa and a simultaneous increase in sperm DNA fragmentation. Based on this pathogenic pathway, it can be hypothesized that SARS-CoV-2 could increase sperm DNA fragmentation, which might affect fertilizing potential. Along the same lines, SARS-CoV-2 may affect oocyte performance through mechanisms that increase oxidative stress.

As SARS-CoV-2 acts through the angiotensin-converting enzyme 2 (ACE2) receptor, this was proposed as an additional pathway affecting ovaria follicles and oocytes. ACE2 receptors are expressed in human ovaries, while angiotensin has been detected in measurable amounts in the follicular fluid . Therefore, a possible negative impact of the virus through an interaction between the oocyte and the somatic cells cannot be ruled out.

The COVID-19 pandemic exerted tremendous pressure on scientists to develop safe and effective vaccines. A few delivery systems for next-generation vaccines against COVID-19 were introduced. The new-generation vaccines include only a specific antigen or antigens of the pathogen, instead of the whole pathogen, thus providing a better safety profile. While SARS-CoV-2 has four main structural proteins, the spike protein (S) which is located at the outer surface of the virus particles and can bind to ACE2 on the cell surface and causes receptor-mediated endocytosis of the virus, is the main target to evoke the self-immune system.

The mRNA vaccines represent the newest generation of vaccines in which all components can be engineered via chemical synthesis. Due to the mRNA molecules' low apparent transfection efficacy, lipid nanoparticles (LNPs) are often used to incorporate the mRNA molecules for transfection purposes. An additional advantage of the mRNA vaccine is that the antigen expression generated by the mRNA is a transient process and therefore the risk of host DNA integration is negligible. Furthermore, elimination of live materials poses an advantage from a quality control standpoint and allows quick product switching in manufacturing facilities. Since the process is fully-synthetic it also eliminates the risk of disease transmissions from the manufacturing facility. The effect of the systemic generation and introduction of just the S protein of the SARS-CoV-2 could have a negative influence on ovarian follicles and oocytes has not been studied yet.

Anti Mullarian Hormone (AMH) is a glycoprotein produced by the granulosa cells of the antral follicles. Its circulating levels are associated with the fertility state of the ovary and in contrast to other hormones are not influenced by the state of the menstrual cycle. Therefore, AMH levels are considered the measurement of choice for estimating ovarian reserve.

As Israel is the first country to widely vaccinate its population using the mRNA vaccines and due to all the aforementioned, the aim of this study is to evaluate the influence of the mRNA vaccines on ovarian reserve estimated by the change in AMH before and three-month following vaccination.

Material and Methods:

This is a prospective study including females that are planning to be vaccinated in Israel. Women will be asked to sign an informed consent to participate in the study while visiting the ambulatory vaccinating clinics before being vaccinated. Medical information will be collected by the research team during this visit using computerized questionnaire. Blood samples will be collected for AMH analysis before administration of the first mRNA vaccine shot. A follow up visit will be scheduled at three months after the first vaccination. During this visit, blood samples will be collected for AMH levels and for anti Covid-19 antibody levels (Serology). Additionally, women will be asked to complete a second computerized questionnaire which focused on possible adverse effects following vaccinations and gynecological well-being at 3,6 and 12 months from recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Age 11-42
* No previous exposure to Covid-19 vaccine (first or second dose)
* No known past Covid-19 infection

Exclusion Criteria:

* Premature ovarian failure
* Pregnancy
* Fertility treatment
* Past Covid-19 infection

Ages: 11 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Women in reproductive age
Study Population: Females (age 11 to 42) that are planning to be vaccinated in Israel
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Delta in AMH levels | From first vaccination until the second AMH sampling - after three month
  AMA levels on recruitment minos AMH levels after three months

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided
On request

REFERENCES:
- [Result] Anifandis G, Messini CI, Daponte A, Messinis IE. COVID-19 and fertility: a virtual reality. Reprod Biomed Online. 2020 Aug;41(2):157-159. doi: 10.1016/j.rbmo.2020.05.001. Epub 2020 May 8. PMID 32466995
- [Result] Joguet G, Mansuy JM, Matusali G, Hamdi S, Walschaerts M, Pavili L, Guyomard S, Prisant N, Lamarre P, Dejucq-Rainsford N, Pasquier C, Bujan L. Effect of acute Zika virus infection on sperm and virus clearance in body fluids: a prospective observational study. Lancet Infect Dis. 2017 Nov;17(11):1200-1208. doi: 10.1016/S1473-3099(17)30444-9. Epub 2017 Aug 23. PMID 28838639
- [Result] Percivalle E, Zavattoni M, Fausto F, Rovida F. Zika virus isolation from semen. New Microbiol. 2017 Jul;40(3):197-198. Epub 2017 May 17. PMID 28513814
- [Result] Khomich OA, Kochetkov SN, Bartosch B, Ivanov AV. Redox Biology of Respiratory Viral Infections. Viruses. 2018 Jul 26;10(8):392. doi: 10.3390/v10080392. PMID 30049972
- [Result] Liu M, Chen F, Liu T, Chen F, Liu S, Yang J. The role of oxidative stress in influenza virus infection. Microbes Infect. 2017 Dec;19(12):580-586. doi: 10.1016/j.micinf.2017.08.008. Epub 2017 Sep 14. PMID 28918004
- [Result] Agarwal A, Rana M, Qiu E, AlBunni H, Bui AD, Henkel R. Role of oxidative stress, infection and inflammation in male infertility. Andrologia. 2018 Dec;50(11):e13126. doi: 10.1111/and.13126. PMID 30569652
- [Result] Dutta S, Majzoub A, Agarwal A. Oxidative stress and sperm function: A systematic review on evaluation and management. Arab J Urol. 2019 Apr 24;17(2):87-97. doi: 10.1080/2090598X.2019.1599624. eCollection 2019. PMID 31285919
- [Result] Homa ST, Vassiliou AM, Stone J, Killeen AP, Dawkins A, Xie J, Gould F, Ramsay JWA. A Comparison Between Two Assays for Measuring Seminal Oxidative Stress and their Relationship with Sperm DNA Fragmentation and Semen Parameters. Genes (Basel). 2019 Mar 19;10(3):236. doi: 10.3390/genes10030236. PMID 30893955
- [Result] Kuhn JH, Li W, Choe H, Farzan M. Angiotensin-converting enzyme 2: a functional receptor for SARS coronavirus. Cell Mol Life Sci. 2004 Nov;61(21):2738-43. doi: 10.1007/s00018-004-4242-5. PMID 15549175
- [Result] Reis FM, Bouissou DR, Pereira VM, Camargos AF, dos Reis AM, Santos RA. Angiotensin-(1-7), its receptor Mas, and the angiotensin-converting enzyme type 2 are expressed in the human ovary. Fertil Steril. 2011 Jan;95(1):176-81. doi: 10.1016/j.fertnstert.2010.06.060. Epub 2010 Aug 1. PMID 20674894
- [Result] Wang J, Peng Y, Xu H, Cui Z, Williams RO 3rd. The COVID-19 Vaccine Race: Challenges and Opportunities in Vaccine Formulation. AAPS PharmSciTech. 2020 Aug 5;21(6):225. doi: 10.1208/s12249-020-01744-7. PMID 32761294
- [Result] Vartak A, Sucheck SJ. Recent Advances in Subunit Vaccine Carriers. Vaccines (Basel). 2016 Apr 19;4(2):12. doi: 10.3390/vaccines4020012. PMID 27104575
- [Derived] Mohr-Sasson A, Haas J, Sivan M, Zehori Y, Hemi R, Orvieto R, Afek A, Rabinovici J. The effects of Covid-19 mRNA vaccine on adolescence gynecological well-being. Arch Gynecol Obstet. 2023 May;307(5):1625-1631. doi: 10.1007/s00404-023-06981-2. Epub 2023 Mar 5. PMID 36871101
- [Derived] Mohr-Sasson A, Haas J, Abuhasira S, Sivan M, Doitch Amdurski H, Dadon T, Blumenfeld S, Derazne E, Hemi R, Orvieto R, Afek A, Rabinovici J. The effect of Covid-19 mRNA vaccine on serum anti-Mullerian hormone levels. Hum Reprod. 2022 Mar 1;37(3):534-541. doi: 10.1093/humrep/deab282. PMID 34935913